CLINICAL TRIAL: NCT02131896
Title: The Effects of Mediterranean Diet on Remission, Lipid Profile, Weight and Body Composition in Children and Adolescents With Newly Diagnosed Type 1 Diabetes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment difficulties
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: rmc7800ctil
Record Dates: First submitted 2014-05-04; First posted 2014-05-06 (Estimated); Last update posted 2017-10-20 (Actual); Status verified 2017-01

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 Diabetes; Newly diagnosed; Lipid profile; Mediterranean diet
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mediterranean Diet (Experimental): Mediterranean Diet
  Interventions: Other: Interventional arm-Mediterranean diet
- Regular nutritional instructions (Active Comparator): Regular nutritional instructions
  Interventions: Other: Control Arm- regular nutritional instructions in accordance with the accepted nutritional guidelines

INTERVENTIONS:
Other: Interventional arm-Mediterranean diet
  Arms: Mediterranean Diet
Other: Control Arm- regular nutritional instructions in accordance with the accepted nutritional guidelines
  Arms: Regular nutritional instructions

SUMMARY:
Nutritional therapy has a major role in diabetes care, achieving and maintaining metabolic control: normal glucose homeostasis, normal lipid profile, normal blood pressure and desirable weight. Controlled nutritional diet, as introduced by the professional committees aims at achieving better general health condition.

There is a growing body of evidence showing that Mediterranean diet has a major role in prevention of diabetes sequelae in type 2 diabetes patients. Hitherto, the effects of Mediterranean diet on patients with type 1 diabetes has not been studied, with the exception of one Italian study.

Six months after education to consume Mediterranean diet in a cohort of 96 children with type 1 diabetes the authors observed decreased fat and cholesterol consumption, increased dietary fiber consumption, lower LDL cholesterol levels and better HDL to LDL cholesterol ratio.

The proposed study is aimed to assess the impact of Mediterranean nutrition compared to the accepted nutritional guidelines, in newly diagnosed type 1 children and adolescents on lipid profile, metabolic control, C peptide, daily insulin dose, Inflammatory parameters, endothelial function and anthropometric parameters 12 months following diagnosis.

The study designed as a two parallel arms, randomized, single center, intervention study.

Patients enrolled to the study will be randomly assigned, to one of the following groups in a 1:1 ratio. Interventional Arm: Patients assigned to the interventional arm will receive nutritional instructions of Mediterranean diet and Control Group: Patients assigned to the interventional arm will receive regular nutritional instructions in accordance with the accepted nutritional guidelines

ELIGIBILITY:
Inclusion Criteria:

* Parents/guardian are willing and able to sign an informed consent form
* Age 5-18 years
* Diagnosis with type 1 diabetes for up to 2 months prior to screening
* Peak C peptide > o.2 pmol/mL

Exclusion Criteria:

* The patient has any significant disease or conditions, including psychiatric disorders that in the opinion of the principal investigator might interfere with patient's compliance or ability to complete the study
* Any concomitant disease that might impact body composition, physical activity level and/or eating habits
* Active celiac disease, hashimoto thyroiditis or uncontrolled Graves' disease
* Down syndrome, Turner, inflammatory bowel disease
* Patients treated with antipsychotic drugs, steroids, or other drugs that might affect body weight and appetite.
* Patient who suffers from eating disorders
* Patients participating in other device or drug studies

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2014-12-01 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
lipid profile | At the end of the study-after 12 months
  fasting blood lipid profile

SECONDARY OUTCOMES:
Metabolic control | At the end of the study-after 12 months
  Metabolic control expressed as HbA1c level
mean and SD of blood glucose | At the end of the study-after 12 months
  Metabolic control expressed as mean and SD of downloaded blood glucose values from patient's personal glucometer
Peak stimulated C peptide | At the end of the study- after 12 months
  Peak stimulated C peptide > o.2 pmol/mL
Daily insulin dose | At the end of the study- after 12 months
  Daily insulin dose adjusted for body weight
Percent of subjects who require a daily insulin dose < o,5 IU/kg | At the end of the study- after 12 months
Frequency and severity of hypoglycemic episodes | At the end of the study- after 12 months
Anthropometric parameters | At the end of the study- after 12 months
  Anthropometric parameters: Body weight ,BMI SDS, body composition and weight change from diagnosis to 12 months after diagnosis
weight change from at least 1 year before diagnosis to 12 months after diagnosis | At the end of the study-after 12 months
Inflammatory parameters | At the end of the study-after 12 months
  Inflammatory parameters: TNF, CRP, IL-6, fibrinogen
Endothelial function | At the end of the study-after 12 months
  Endothelial function: Doppler assessment of the tunica intima

CONTACTS AND LOCATIONS:
Overall Officials: Liat de Vries, Dr, Principal Investigator — Schneider Children's Medical Center
Locations (1):
- Schneider Children's Medical Center, Petah Tikva, Israel